CLINICAL TRIAL: NCT05107882
Title: Retinal Deep PhenotypingTM Platform for Cerebral Amyloid Status Evaluation: a Validation Study
Brief Title: Optina Diagnostics' Cerebral ß-Amyloid Status (CAS) Test
Acronym: REPHRASE
Status: Completed | Type: Observational
Sponsor: Optina Diagnostics Inc. (Industry)
Collaborators: Eastern Virginia Medical School (Other); The Cleveland Clinic (Other); University of Washington (Other); Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DOC100464
Record Dates: First submitted 2021-10-21; First posted 2021-11-04 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational, cross-sectional study is designed to validate a novel diagnostic test for the detection of phenotypic changes in the retina that correlate with likely PET amyloid status (negative or positive), to aid in the evaluation of adult patients with cognitive impairment who are being evaluated for Alzheimer's disease and other causes of cognitive decline. The CAS test is an adjunct to other diagnostic evaluations, and is indicated for use with the Optina Diagnostics' MHRC (K200254).

DETAILED DESCRIPTION:
This non-interventional, cross-sectional study is designed to validate a novel diagnostic test, the Optina Diagnostics' Cerebral ß-Amyloid Status (CAS) test, for the detection of phenotypic changes in the retina that correlate with likely PET amyloid status (positive or negative). The CAS test is an adjunct to other diagnostic evaluations, and is indicated for use with the Optina Diagnostics' MHRC for imaging the retina. The study objective is to characterize the performance of the diagnostic CAS test in the target population of adult patients fifty (50) years and older with cognitive impairment, who are being evaluated for Alzheimer's disease (AD) and other causes of cognitive decline. The data generated in this study will provide evidence to be used in the assessment of the benefits and risks associated with use of the device in the intended population. The primary endpoint is to demonstrate accuracy of the Optina Diagnostics' CAS test compared to amyloid-PET status, as determined by a majority of three (3) qualified, independent PET Readers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 50 years and older (inclusive).
* Individuals with reported cognitive complaint (self or from an informant) under clinical investigation by a health professional for cognitive impairment where Alzheimer's disease (AD) is one of the differential diagnoses.
* Demonstrated cognitive impairment as evidenced by at least one of the following:

  1. Mini Mental State Examination (MMSE) score < 26/30
  2. Montreal Cognitive Assessment (MoCA) score < 26/30
  3. Score > 1 Standard Deviation below population mean on a standardized neuropsychological test (in any domain), based on normative data from age-, sex-, education-, and where possible, race-matched peers [Based on guidelines for detecting Mild Cognitive Impairment due to AD (Albert et al., 2011)]
* Clinical laboratory assessment (complete blood count [CBC], standard blood chemistry profile, thyroid stimulating hormone [TSH], vitamin B12) within the 6 months prior to enrollment.
* Cognitive impairment on the above test/s is unable to be fully explained by systemic, neurological or psychiatric disorders other than Alzheimer's disease.
* Capacity to give informed consent by patient or substitute decision maker.
* Ability to undergo PET and MRI scans.

Exclusion Criteria:

* Any ophthalmologic condition that would prevent obtaining retinal imaging and/or could interfere with the analysis of the MHRC images by the CAS, including:

  1. Pupil dilation contraindicated (due to a pathology, or presence of 3 quadrants with Van Herick grading of 0 or 1 without iridotomy)
  2. Inadequate pupil dilatation (< 6mm diameter) preventing uniform illumination of the retina with the MHRC
  3. Diagnosis of glaucoma or signs of glaucoma (excavation ratio ≥0.7)
  4. Signs of vascular occlusion or retinopathy (microaneurysm, exudate, hemorrhage or edema) within a diameter of 10 mm from the mid-point between the optic nerve head and the macula
  5. Presence of drusen and/or age-related macular degeneration (AREDS 9-step scale ≥4 - cumulative drusen area diameter ≥ 250 um, pigmentary changes and cumulative drusen area diameter ≥ 63 um or pigmentary changes and cumulative geographic atrophy area diameter ≥ 354 um)
  6. Macular anomaly (e.g., macular hole, dystrophy, degeneration)
  7. Nuclear sclerosis > 2 (LOCS II four-point grading system) or presence of central cortical or central posterior subcapsular cataract
  8. Refractive error outside the range of -15 D to +15 D
  9. Scar, atrophy, naevus, tumor, eepiretinal membrane or retinal pucker with a cumulative area > 1 disc area within a diameter of 10 mm from the mid-point between the optic nerve head and the macula
  10. Papilledema
  11. Deficient visual fixation (inability to fixate for at least 2 s)
  12. Corneal or media opacities (e.g., Weiss ring) affecting retinal imaging on a cumulative area > 1 disc area within a diameter of 10 mm from the mid-point between the optic nerve head and the macula (i.e., the area of interest for the MHRC imaging)
* Inability of obtaining at least 3 images of satisfactory quality with the MHRC per the Optina Diagnostics quality index software and /or per the eye specialists' evaluation.
* Impossibility of obtaining a satisfactory quality amyloid-PET scan for interpretation by imaging specialists.
* Individuals who currently or have previously taken cerebral amyloid modifying medication.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population for the Optina Diagnostics' CAS test is men and women 50 years and older who are under clinical investigation for cognitive impairment where Alzheimer's disease (AD) is one of the possible differential diagnoses.
  As concomitant eye pathologies or conditions could interfere with CAS algorithm, individuals with certain ocular pathologies or conditions, including glaucoma, age-related macular degeneration (AMD), retinopathies, and advanced cataracts, will not be included in the target population at this time. Work is on-going to improve the CAS classifier algorithm with the goal to include these individuals in the target population at a later date.
Sampling Method: Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Retinal beta-amyloid detection | 1 year
  Presence of absence of beta-amyloid plaques in the retina where the accuracy will be assessed using positive percent agreement (PPA) and negative percent agreement (NPA) with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Okhravi, MD, PhD FRPC, Principal Investigator — Eastern Virginia Medical Center; Richard Bergeron, PhD FRPC, Principal Investigator — Ottawa Memory Clinic and Clinic Memoire Outaouais; Suman Jayadev, MD, Principal Investigator — University of Washington; Charles Bernick, MD, MPH, Principal Investigator — Cleveland Clinic Lou Ruvo Center for Brain; Sandra Black, MD, Principal Investigator — Sunnybrook Research Institute (SRI); Jorge P. Bruno, MD, Principal Investigator — Ezy Medical Research; Giovanni J Marotta, MD, FRCP(C), Principal Investigator — Centricity Research
Locations (7):
- United States (4):
  - Ezy Medical Research, Miami, Florida
  - Lou Ruvo Center for Brain Health at Cleveland Clinic (LR-CC), Las Vegas, Nevada
  - East Virginia Medical School (EVMS), Norfolk, Virginia
  - University of Washington (MBWC), Seattle, Washington
- Canada (3):
  - Ottawa Memory Clinic (OMC), Ottawa, Ontario
  - Centricity Research, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No